CLINICAL TRIAL: NCT01238991
Title: A Phase Iia, Multicenter, Treatment Assigned, Open-label, Long-term Extension Study To Determine Safety, Tolerability, And Immunogenicity Of Acc-001 With Qs-21 Adjuvant In Japanese Subjects With Mild To Moderate Alzheimer's Disease
Brief Title: Long Term Extension Study Evaluating Safety, Tolerability And Immunogenicity Of ACC-001 In Japanese Subjects With Mild To Moderate Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: JANSSEN Alzheimer Immunotherapy Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2571001; 3134K1-2207 (Other: Alias Study Number)
Record Dates: First submitted 2010-10-21; First posted 2010-11-11 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2014-12-22 (Estimated); Status verified 2014-12

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — vanutide cridificar

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ACC-001 (3 micrograms) + QS-21 (Experimental): Active vaccine dose of 3 micrograms +adjuvant, IM injection, at Day 1, month 6, 12 and 18
  Interventions: Biological: ACC-001
- ACC-001 (10 micrograms) + QS-21 (Experimental): Active vaccine dose of 10 micrograms +adjuvant, IM injection, at Day 1, month 6, 12 and 18
  Interventions: Biological: ACC-001
- ACC-001 (30 micrograms) + QS-21 (Experimental): Active vaccine dose of 30 micrograms +adjuvant, IM injection, at Day 1, month 6, 12 and 18
  Interventions: Biological: ACC-001

INTERVENTIONS:
Biological: ACC-001 — IM injection, dose of 3 micrograms, at Day 1, month 6, 12 and 18
  Arms: ACC-001 (3 micrograms) + QS-21
Biological: ACC-001 — IM injection, dose of 10 micrograms, at Day 1, month 6, 12 and 18
  Arms: ACC-001 (10 micrograms) + QS-21
Biological: ACC-001 — IM injection, dose of 30 micrograms, at Day 1, month 6, 12 and 18
  Arms: ACC-001 (30 micrograms) + QS-21

SUMMARY:
The purpose of this long term extension study is to assess safety, tolerability and immunogenicity of ACC-001 with QS-21 adjuvant in Japanese subjects with mild to moderate AD who were randomized in the preceding P2 double blind studies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects randomized under previous 3134K1-2202-JA (NCT00752232) and 3134K1-2206-JA (NCT00959192) and met all inclusion criteria and non of the exclusion criteria.
* Screening brain MRI scan is consistent with the diagnosis of AD.
* MMSE score 10 and above.

Exclusion Criteria:

* Significant neurological diseases other than AD.
* Brain MRI evidence of vasogenic edema during the preceding studies.
* Clinically significant illness.

Ages: 52 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- Japan (11):
  - Meitetsu Hospital, Nagoya, Aichi-ken
  - Ibaraki Prefectural Central Hospital, Kasama, Ibaraki
  - Shonan Atsugi Hospital, Atsugi, Kanagawa
  - Kitasato University East Hospital, Sagamihara-shi, Kanagawa
  - Suwa Red Cross Hospital, Suwa, Nagano
  - Tazuke Kofukai Medical Research Institute Kitano Hospital, Osaka, Osaka
  - Osaka Medical College Hospital, Takatsuki, Osaka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Juntendo Tokyo Koto Geriatric Medical Center, Koto-ku, Tokyo
  - The Tokyo Jikei University School of Medicine, Minato-ku, Tokyo
  - Kanto Central Hospital of the Mutual Aid Association of Public School Teachers, Setagaya-ku, Tokyo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2571001&StudyName=Long%20Term%20Extension%20Study%20Evaluating%20Safety%2C%20Tolerability%20And%20Immunogenicity%20Of%20ACC-001%20In%20Japanese%20Subjects%20With%20Mild%20To%20Moderate%20Alzhe

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study enrolled those who completed the preceding studies (NCT00752232 and NCT00959192), where active vaccine ACC-001 (3, 10 or 30 μg) + adjuvant QS-21 (50 μg), as well as ACC-001, QS-21 and phosphate buffered saline (PBS) alone, were administered at Day 1, month 3, 6, 9 and 12 and at Day 1, month 1, 3, 6 and 12, respectively.
Groups:
- 3 μg ACC-001+QS-21: A group of participants who received intramuscular (IM) injection of active vaccine ACC-001 (3 μg) + adjuvant QS-21 (50 μg) both in the preceding studies and in this study (Day 1, month 6, 12, and 18)
- QS-21+(3 μg ACC-001+QS-21): A group of participants who received IM injection of adjuvant QS-21 (50 μg) in the preceding studies and active vaccine ACC-001 (3 μg) + adjuvant QS-21 (50 μg) in this study (Day 1, month 6, 12, and 18)
- 10 μg ACC-001+QS-21: A group of participants who received IM injection of active vaccine ACC-001(10 μg) + adjuvant QS-21 (50 μg) both in the preceding studies and in this study (Day 1, month 6, 12, and 18)
- 10 μg ACC-001+ (10 μg ACC-001+QS-21): A group of participants who received IM injection of active vaccine ACC-001(10 μg) in the preceding studies and ACC-001 (10 μg) + adjuvant QS-21 (50 μg) in this study (Day 1, month 6, 12, and 18)
- QS-21+(10 μg ACC-001+QS-21): A group of participants who received IM injection of adjuvant QS-21 (50 μg) in the preceding studies and active vaccine ACC-001(10 μg) + adjuvant QS-21 (50 μg) in this study (Day 1, month 6, 12, and 18)
- PBS+(10 μg ACC-001+QS-21): A group of participants who received IM injection of PBS in the preceding studies and active vaccine ACC-001 (10 μg) + adjuvant QS-21 (50 μg) in this study (Day 1, month 6, 12, and 18)
- 30 μg ACC-001+QS-21: A group of participants who received IM injection of active vaccine ACC-001 (30 μg) + adjuvant QS-21 (50 μg) both in the preceding studies and in this study (Day 1, month 6, 12, and 18)
- 30 μg ACC-001+(30 μg ACC-001+QS-21): A group of participants who received IM injection of active vaccine ACC-001(30 μg) in the preceding studies and ACC-001(30 μg) + adjuvant QS-21 (50 μg) in this study (Day 1, month 6, 12, and 18)
- QS-21+(30 μg ACC-001+QS-21): A group of participants who received IM injection of adjuvant QS-21 (50 μg) in the preceding studies and active vaccine ACC-001(30 μg) + adjuvant QS-21 (50 μg) in this study (Day 1, month 6, 12, and 18)
- PBS+(30 μg ACC-001+QS-21): A group of participants who received IM injection of PBS in the preceding studies and active vaccine ACC-001(30 μg) + adjuvant QS-21 (50 μg) in this study (Day 1, month 6, 12, and 18)
Period: Overall Study
Arm/Group | 3 μg ACC-001+QS-21 | QS-21+(3 μg ACC-001+QS-21) | 10 μg ACC-001+QS-21 | 10 μg ACC-001+ (10 μg ACC-001+QS-21) | QS-21+(10 μg ACC-001+QS-21) | PBS+(10 μg ACC-001+QS-21) | 30 μg ACC-001+QS-21 | 30 μg ACC-001+(30 μg ACC-001+QS-21) | QS-21+(30 μg ACC-001+QS-21) | PBS+(30 μg ACC-001+QS-21)
Started | 7 | 3 | 11 | 6 | 5 | 2 | 8 | 5 | 4 | 2
Received Treatment | 7 | 3 | 11 | 6 | 5 | 2 | 8 | 5 | 4 | 2
Completed | 5 | 3 | 5 | 4 | 3 | 2 | 0 | 0 | 0 | 0
Not Completed | 2 | 0 | 6 | 2 | 2 | 0 | 8 | 5 | 4 | 2
Not completed — Adverse Event | 1 | 0 | 3 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 4 | 2 | 2
Not completed — Caregiver's request | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Admission to a nursing home | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 3 μg ACC-001+QS-21: A group of participants who received IM injection of active vaccine ACC-001 (3 μg) + adjuvant QS-21 (50 μg) both in the preceding studies and in this study (Day 1, month 6, 12, and 18)
- Total: Total of all reporting groups
Arm/Group | 3 μg ACC-001+QS-21 | QS-21+(3 μg ACC-001+QS-21) | 10 μg ACC-001+QS-21 | 10 μg ACC-001+ (10 μg ACC-001+QS-21) | QS-21+(10 μg ACC-001+QS-21) | PBS+(10 μg ACC-001+QS-21) | 30 μg ACC-001+QS-21 | 30 μg ACC-001+(30 μg ACC-001+QS-21) | QS-21+(30 μg ACC-001+QS-21) | PBS+(30 μg ACC-001+QS-21) | Total
Number analyzed (Participants) | 7 | 3 | 11 | 6 | 5 | 2 | 8 | 5 | 4 | 2 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (9.8) | 73.3 (9.2) | 67.5 (9.8) | 69.5 (6.9) | 65.2 (6.7) | 70.5 (7.8) | 73.9 (5.4) | 71.2 (2) | 64 (7.1) | 68.5 (2.1) | 69.2 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 8 | 4 | 3 | 2 | 4 | 3 | 4 | 1 | 36
  Male | 3 | 0 | 3 | 2 | 2 | 0 | 4 | 2 | 0 | 1 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Emergent Adverse Events (AEs) by Severity
Description: Number of mild, moderate, and severe AEs (mild = does not interfere with subject's usual function; moderate = interferes to some extent with subject's usual function; severe = interferes significantly with subject's usual function)
Time Frame: Baseline up to 24 months
Population: The population for safety analysis consisted of all enrolled participants who received at least one injection of study medication in this study.
Measure: Number; unit: Events
Groups:
- 3 μg ACC-001 Treat: A group of participants who received IM injection of active vaccine ACC-001 (3 μg) + adjuvant QS-21 (50 μg) both in the preceding studies and in this study (Day 1, month 6, 12, and 18)
- 3 μg Control: A group of participants who received IM injection of adjuvant QS-21 (50 μg) in the preceding studies and active vaccine ACC-001 (3 μg) + adjuvant QS-21 (50 μg) in this study (Day 1, month 6, 12, and 18)
- 10 μg ACC-001 Treat: A group of participants who received IM injection of active vaccine ACC-001(10 μg) with or without adjuvant QS-21 (50 μg) in the preceding studies and ACC-001 (10 μg) + adjuvant QS-21 (50 μg) in this study (Day 1, month 6, 12, and 18)
- 10 μg Control: A group of participants who received IM injection of adjuvant QS-21 (50 μg) or PBS in the preceding studies and active vaccine ACC-001(10 μg) + adjuvant QS-21 (50 μg) in this study (Day 1, month 6, 12, and 18)
- 30 μg ACC-001 Treat: A group of participants who received IM injection of active vaccine ACC-001 (30 μg) with or without adjuvant QS-21 (50 μg) in the preceding studies and ACC-001 (30 μg) + adjuvant QS-21 (50 μg) in this study (Day 1, month 6, 12, and 18)
- 30 μg Control: A group of participants who received IM injection of adjuvant QS-21 (50 μg) or PBS in the preceding studies and active vaccine ACC-001 (30 μg) + adjuvant QS-21 (50 μg) in this study (Day 1, month 6, 12, and 18)
Arm/Group | 3 μg ACC-001 Treat | 3 μg Control | 10 μg ACC-001 Treat | 10 μg Control | 30 μg ACC-001 Treat | 30 μg Control
Number analyzed (Participants) | 7 | 3 | 17 | 7 | 13 | 6
Events
  Mild | 14 | 7 | 97 | 38 | 28 | 17
  Moderate | 2 | 0 | 14 | 2 | 3 | 4
  Severe | 0 | 0 | 6 | 0 | 2 | 0

2. Primary Outcome: Number of Participants With Brain Abnormalities in Magnetic Resonance Imaging (MRI) Data
Description: Number of participants with brain abnormalities in MRI data that are either consistent or not consistent with AD, as determined by radiologists.
Time Frame: Baseline up to 24 months
Population: The population for safety analysis consisted of all enrolled participants who received at least one injection of study medication in this study. Since the study was early terminated and the data could not be obtained as planned, the MRI data were not summarized.
Arm/Group | 3 μg ACC-001 Treat | 3 μg Control | 10 μg ACC-001 Treat | 10 μg Control | 30 μg ACC-001 Treat | 30 μg Control
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Abnormalities in Neurological Examination
Description: Number of participants with abnormalities in neurological examinations as determined by the investigators. Neurological examinations included Mental Status, Speech, Cranial Nerve Function, Cranial Nerve II, Sensory Function, Motor Function, Coordination, Gait and Station, Reflexes and Deep Tendon Reflexes.
Time Frame: Baseline of the preceding studies through 24 months of this study
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | 3 μg ACC-001 Treat | 3 μg Control | 10 μg ACC-001 Treat | 10 μg Control | 30 μg ACC-001 Treat | 30 μg Control
Number analyzed (Participants) | 7 | 3 | 17 | 7 | 13 | 6
Participants
  Mental Status | 0 | 0 | 2 | 0 | 0 | 1
  Speech | 0 | 0 | 1 | 0 | 0 | 0
  Cranial Nerve Function | 0 | 0 | 0 | 0 | 0 | 0
  Cranial Nerve II | 0 | 0 | 1 | 0 | 0 | 0
  Sensory Function | 0 | 0 | 0 | 0 | 0 | 1
  Motor Function | 0 | 0 | 0 | 0 | 0 | 0
  Coordination | 0 | 0 | 0 | 0 | 0 | 0
  Gait and Station | 0 | 0 | 2 | 0 | 1 | 0
  Reflexes | 0 | 0 | 0 | 0 | 0 | 0
  Deep Tendon Reflexes | 0 | 0 | 0 | 0 | 0 | 0

4. Other Pre Specified Outcome: Anti-A-beta IgG (Immunoglobulin G) Titer at Specified Visits
Description: Geometric mean of anti-a-beta IgG titer from baseline of the preceding studies through the end of this study
Time Frame: Baseline of preceding studies to month 24 of this study (Week 210)
Population: The immunogenicity analysis population consisted of those in the safety analysis population who had baseline immunogenicity evaluation in the preceding study and at least one immunogenicity evaluation post injection.
Measure: Geometric Mean (95% Confidence Interval); unit: Units/mL
Groups:
- 10 μg ACC-001+(10 μg ACC-001+QS-21): A group of participants who received IM injection of active vaccine ACC-001 (10 μg) in the preceding studies and ACC-001 (10 μg) + adjuvant QS-21 (50 μg) in this study (Day 1, month 6, 12, and 18)
- PBS+(30 μg ACC-001+QS-21): A group of participants who received IM injection of PBS in the preceding studies and active vaccine ACC-001(30 μg) + adjuvant QS-21(50 μg) in this study (Day 1, month 6, 12, and 18)
Arm/Group | 3 μg ACC-001+QS-21 | QS-21+(3 μg ACC-001+QS-21) | 10 μg ACC-001+QS-21 | 10 μg ACC-001+(10 μg ACC-001+QS-21) | QS-21+(10 μg ACC-001+QS-21) | PBS+(10 μg ACC-001+QS-21) | 30 μg ACC-001+QS-21 | 30 μg ACC-001+(30 μg ACC-001+QS-21) | QS-21+(30 μg ACC-001+QS-21) | PBS+(30 μg ACC-001+QS-21)
Number analyzed (Participants) | 7 | 3 | 11 | 6 | 5 | 2 | 8 | 5 | 4 | 2
Units/mL
  Pre-study (n=7, 3, 11, 6, 5, 2, 8, 5, 4, 2) | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 2 (n=7, 3, 11, 6, 5, 2, 8, 5, 4, 2) | 60.3 [38.1 to 95.5] | 50.0 [50.0 to 50.0] | 67.2 [34.7 to 130.1] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 4 (n=4, 2, 7, 0, 3, 0, 5, 0, 2, 0) | 158.5 [18.2 to 1381.1] | 50.0 [50.0 to 50.0] | 73.5 [36.6 to 147.2] | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | 50.0 [50.0 to 50.0] | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | 50.0 [50.0 to 50.0] | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | 50.0 [50.0 to 50.0] | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week.
  Week 6 (n=7, 3, 11, 6, 5, 2, 8, 5, 4, 2) | 797.2 [49.7 to 12776.7] | 50.0 [50.0 to 50.0] | 1346.8 [289.6 to 6264.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 924.1 [142.2 to 6003.5] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 8 (n=4, 2, 7, 0, 3, 0, 5, 0, 2, 0) | 3202.0 [168.8 to 60744.5] | 50.0 [50.0 to 50.0] | 2950.3 [837.0 to 10399.3] | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | 50.0 [50.0 to 50.0] | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | 2543.1 [969.3 to 6672.1] | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | 50.0 [50.0 to 50.0] | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week.
  Week 10 (n=7, 3, 11, 6, 5, 2, 8, 5, 4, 2) | 494.2 [49.1 to 4970.9] | 50.0 [50.0 to 50.0] | 638.8 [160.2 to 2547.6] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 386.9 [87.7 to 1707.3] | 61.3 [34.9 to 107.6] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 14 (n=7, 3, 11, 6, 5, 2, 8, 5, 4, 2) | 6174.8 [1628.1 to 23419.5] | 50.0 [50.0 to 50.0] | 5696.9 [2541.3 to 12771.2] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 5266.4 [1852.1 to 14975.0] | 207.5 [24.9 to 1726.5] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 16 (n=7, 3, 11, 6, 5, 2, 8, 5, 4, 2) | 4239.5 [895.3 to 20075.3] | 50.0 [50.0 to 50.0] | 3471.2 [1569.0 to 7680.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 5014.4 [1788.3 to 14060.5] | 166.0 [20.3 to 1355.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 24 (n=7, 3, 11, 6, 5, 2, 8, 5, 4, 2) | 1292.4 [263.8 to 6331.1] | 50.0 [50.0 to 50.0] | 1122.5 [502.5 to 2507.3] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 1765.8 [638.5 to 4883.6] | 133.6 [24.5 to 727.2] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 28 (n=7, 3, 11, 6, 5, 2, 8, 5, 4, 2) | 6460.4 [1521.1 to 27438.5] | 50.0 [50.0 to 50.0] | 6712.0 [1862.9 to 24183.8] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 8383.3 [4000.7 to 17566.9] | 471.9 [24.3 to 9181.4] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 30 (n=7, 3, 11, 6, 5, 2, 8, 5, 4, 2) | 4928.0 [1015.9 to 23904.5] | 50.0 [50.0 to 50.0] | 5417.0 [1626.4 to 18042.7] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 7927.9 [4408.1 to 14258.0] | 408.1 [19.8 to 8412.5] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 34 (n=3, 1, 4, 6, 2, 2, 3, 5, 2, 2) | 992.7 [9.5 to 103353.0] | 50.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | 4480.4 [34.4 to 583150.4] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 7851.2 [1669.4 to 36923.6] | 287.4 [21.2 to 3888.4] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 38 (n=3, 1, 4, 6, 2, 2, 3, 5, 2, 2) | 5444.2 [634.1 to 46744.1] | 50.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | 4923.0 [65.7 to 368774.1] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 18040.4 [1536.5 to 211818.5] | 522.7 [30.5 to 8951.6] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 40 (n=7, 3, 11, 6, 5, 2, 8, 5, 4, 2) | 4584.4 [2315.0 to 9078.7] | 50.0 [50.0 to 50.0] | 2639.5 [839.1 to 8302.7] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 4899.8 [1919.8 to 12505.5] | 408.9 [29.2 to 5733.6] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 50 (n=7, 3, 11, 6, 5, 2, 8, 5, 4, 2) | 2153.0 [1108.4 to 4182.2] | 50.0 [50.0 to 50.0] | 1603.8 [528.8 to 4864.7] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 2587.5 [999.3 to 6699.7] | 205.0 [27.1 to 1549.9] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 54 (n=7, 3, 11, 6, 5, 2, 8, 5, 4, 2) | 5374.9 [2019.8 to 14303.3] | 50.0 [50.0 to 50.0] | 7559.6 [2614.6 to 21857.4] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 10900.6 [5915.4 to 20087.3] | 611.2 [72.8 to 5131.5] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 56 (n=7, 3, 11, 6, 5, 2, 8, 5, 4, 2) | 7811.2 [2656.5 to 22968.2] | 50.0 [50.0 to 50.0] | 6204.2 [1855.1 to 20749.6] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 8052.1 [4251.8 to 15249.1] | 458.0 [65.9 to 3180.4] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 66 (n=7, 3, 11, 6, 5, 2, 8, 5, 4, 2) | 4668.7 [1533.4 to 14214.4] | 50.0 [50.0 to 50.0] | 3877.2 [1217.4 to 12347.8] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 3885.1 [1951.3 to 7735.2] | 227.2 [32.6 to 1582.8] | 194.0 [2.6 to 14517.7] | 50.0 [50.0 to 50.0]
  Week 78 (n=7, 3, 11, 6, 5, 2, 8, 5, 4, 2) | 2983.3 [954.1 to 9328.0] | 50.0 [50.0 to 50.0] | 2488.3 [836.1 to 7405.1] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 2272.0 [1192.1 to 4330.1] | 231.0 [34.2 to 1559.2] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 82 (n=4, 2, 11, 6, 5, 2, 8, 5, 4, 2) | 16812.5 [2685.3 to 105259.9] | 50.0 [50.0 to 50.0] | 9783.0 [3283.5 to 29148.1] | 108.7 [41.8 to 282.7] | 110.7 [12.2 to 1006.4] | 50.0 [50.0 to 50.0] | 14160.9 [8518.5 to 23540.4] | 975.6 [209.4 to 4546.5] | 196.4 [30.3 to 1275.0] | 385.1 [0.0 to 70941268874642]
  Week 84 (n=4, 2, 11, 6, 5, 2, 8, 5, 4, 2) | 14763.7 [3422.9 to 63679.1] | 188.0 [188.0 to 188.0] | 7058.6 [2484.5 to 20054.3] | 94.9 [43.4 to 207.3] | 136.0 [18.7 to 989.2] | 109.3 [0.0 to 2265473.2] | 9998.6 [5487.3 to 18218.7] | 768.3 [126.4 to 4669.5] | 383.9 [39.8 to 3700.8] | 316.9 [0.0 to 4897026295844.7]
  Week 91 (n=3, 1, 0, 0, 0, 0, 0, 0, 0, 0) | 1030.3 [51.7 to 20540.2] | 50.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week.
  Week 92 (n=4, 2, 11, 6, 5, 2, 8, 5, 4, 2) | 6100.2 [1730.5 to 21504.2] | 277.1 [1.1 to 71502.3] | 4142.3 [1719.9 to 9976.6] | 67.6 [41.1 to 111.1] | 169.3 [50.3 to 569.9] | 50.0 [50.0 to 50.0] | 4291.7 [2472.4 to 7449.7] | 391.5 [56.2 to 2724.4] | 299.8 [40.3 to 2229.5] | 285.8 [0.0 to 1192613970596.0]
  Week 104 (n=7, 3, 11, 6, 5, 2, 7, 4, 3, 2) | 2173.6 [652.1 to 7244.7] | 83.4 [9.2 to 753.5] | 2224.8 [934.8 to 5295.0] | 50.0 [50.0 to 50.0] | 105.9 [40.1 to 279.5] | 50.0 [50.0 to 50.0] | 3167.0 [1460.6 to 6867.2] | 464.0 [40.3 to 5344.9] | 256.1 [7.6 to 8678.4] | 213.8 [0.0 to 22254714647.2]
  Week 108 (n=7, 3, 11, 6, 5, 2, 7, 4, 4, 2) | 14800.8 [4544.9 to 48199.8] | 872.2 [1.7 to 459286.2] | 8306.6 [4126.8 to 16719.9] | 688.8 [118.8 to 3993.8] | 4818.1 [1026.0 to 22626.7] | 1172.0 [0.0 to 54658314329.3] | 13370.6 [6739.1 to 26527.7] | 3596.0 [469.5 to 26042.1] | 448.0 [4.4 to 45743.6] | 14665.8 [0.0 to 2439205485421.2]
  Week 110 (n=7, 3, 10, 6, 5, 2, 7, 4, 2, 2) | 9185.4 [3237.8 to 26058.4] | 1257.0 [15.9 to 99324.4] | 8081.4 [4125.7 to 15829.8] | 551.4 [81.2 to 3743.4] | 3726.2 [1084.8 to 12799.5] | 497.9 [0.0 to 39348525251.6] | 12209.4 [6421.3 to 23215.2] | 2504.2 [464.4 to 13505.3] | 2670.5 [0.0 to 463269086196.1] | 9454.1 [0.0 to 2972501787380.5]
  Week 116 (n=4, 2, 10, 4, 5, 2, 7, 4, 2, 2) | 1682.2 [38.5 to 73591.4] | 1548.4 [1.3 to 1837780.1] | 5926.3 [2682.3 to 13093.5] | 831.0 [59.8 to 11548.2] | 2335.3 [715.0 to 7628.0] | 258.0 [0.0 to 292460133977.7] | 8613.4 [4540.7 to 16339.2] | 1136.1 [153.1 to 8429.8] | 2929.2 [0.0 to 4137410775629.6] | 5735.6 [0.0 to 50649360975.1]
  Week 118 (n=3, 1, 0, 0, 0, 0, 0, 0, 0, 0) | 4506.7 [59.6 to 340984.3] | 50.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week.
  Week 130 (n=6, 3, 10, 5, 5, 2, 7, 4, 2, 2) | 3312.9 [918.1 to 11954.2] | 323.7 [4.0 to 25932.8] | 2251.0 [704.2 to 7195.9] | 435.9 [45.5 to 4172.4] | 1231.0 [471.1 to 3216.5] | 185.1 [0.0 to 3083418082.5] | 4197.4 [2224.2 to 7921.3] | 516.8 [42.1 to 6345.2] | 1427.2 [0.0 to 61098419244.5] | 3359.9 [0.0 to 416391434.9]
  Week 134 (n=5, 3, 8, 4, 5, 2, 6, 4, 1, 2) | 5904.2 [2760.4 to 12628.6] | 4418.8 [32.8 to 595262.2] | 11064.6 [3340.9 to 36644.9] | 2718.6 [83.6 to 88360.8] | 5233.2 [2190.3 to 12503.5] | 4957.3 [0.0 to 89132252682601] | 6043.9 [1405.3 to 25993.5] | 2189.8 [39.4 to 121572.0] | 4629.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | 14525.7 [1101.4 to 191573.6]
  Week 136 (n=6, 3, 8, 4, 5, 2, 2, 4, 0, 2) | 7816.8 [2323.1 to 26302.4] | 3706.5 [28.6 to 480359.1] | 10195.4 [3243.3 to 32049.6] | 2572.6 [101.9 to 64964.0] | 4614.4 [1945.0 to 10947.8] | 3490.4 [0.0 to 129808983536252] | 18653.9 [20.0 to 17387177.2] | 1799.7 [40.1 to 80796.0] | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | 6296.3 [3108.1 to 12754.9]
  Week 142 (n=3, 1, 0, 0, 0, 0, 0, 0, 0, 0) | 2353.6 [164.1 to 33761.9] | 12571.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week.
  Week 146 (n=3, 2, 9, 4, 5, 2, 2, 4, 0, 2) | 6813.3 [1976.2 to 23490.5] | 979.6 [447.2 to 2146.1] | 7269.6 [2546.0 to 20756.9] | 3252.9 [156.4 to 67657.2] | 3163.7 [1153.6 to 8676.4] | 1338.7 [0.0 to 2432477307830.6] | 9664.4 [6383.5 to 14631.5] | 1022.4 [41.4 to 25279.5] | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | 4277.9 [538.3 to 33999.7]
  Week 156 (n=6, 3, 8, 4, 4, 2, 2, 4, 0, 2) | 2998.5 [853.4 to 10536.3] | 1410.5 [237.4 to 8381.7] | 4600.8 [1798.3 to 11770.3] | 2532.8 [97.0 to 66111.6] | 2880.8 [1242.7 to 6678.3] | 737.9 [0.0 to 11966762355531] | 6706.3 [164.9 to 272699.3] | 706.6 [41.7 to 11981.1] | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | 2643.6 [1902.1 to 3674.2]
  Week 160 (n=5, 3, 7, 4, 2, 2, 1, 2, 0, 1) | 6305.4 [2243.7 to 17719.5] | 1833.3 [101.1 to 33260.5] | 6945.3 [3865.8 to 12477.7] | 4810.2 [366.0 to 63211.9] | 4080.8 [0.0 to 11159747036.1] | 3632.1 [434.2 to 30382.4] | 7731.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | 1779.5 [362.3 to 8741.0] | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | 2518.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable.
  Week 162 (n=6, 3, 8, 4, 4, 2, 0, 0, 0, 0) | 8513.5 [2074.4 to 34940.7] | 1586.1 [125.6 to 20025.2] | 10450.4 [5734.0 to 19046.0] | 6398.1 [417.4 to 98070.7] | 6453.5 [1202.3 to 34641.3] | 2362.8 [0.4 to 13656178.6] | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week.
  Week 171 (n=3, 2, 7, 4, 4, 2, 0, 0, 0, 0) | 8602.3 [4440.7 to 16664.0] | 739.7 [32.9 to 16622.6] | 7551.2 [3117.9 to 18288.2] | 7027.0 [485.8 to 101644.6] | 4351.5 [1055.3 to 17944.0] | 1404.9 [0.0 to 328577560.1] | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week.
  Week 172 (n=2, 1, 0, 0, 0, 0, 0, 0, 0, 0) | 1074.9 [0.1 to 8576667.2] | 2981.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week.
  Week 182 (n=3, 1, 0, 0, 0, 0, 0, 0, 0, 0) | 1944.9 [81.6 to 46329.0] | 2555.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week.
  Week 184 (n=3, 2, 6, 4, 3, 2, 0, 0, 0, 0) | 7062.8 [5311.4 to 9391.7] | 636.6 [4.1 to 98882.9] | 3378.1 [1687.3 to 6763.1] | 5682.1 [345.0 to 93583.6] | 5064.1 [3850.7 to 6659.9] | 824.3 [0.0 to 32731187354.9] | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week.
  Week 186 (n=2, 1, 0, 0, 0, 0, 0, 0, 0, 0) | 3653.9 [0.0 to 8947070499.4] | 13166.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week.
  Week 188 (n=2, 1, 0, 0, 0, 0, 0, 0, 0, 0) | 3033.0 [0.0 to 11447766146.8] | 14096.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week.
  Week 197 (n=3 1, 0, 0, 0, 0, 0, 0, 0, 0) | 2074.7 [78.6 to 54786.4] | 5502.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week.
  Week 210 (n=2, 1, 0, 0, 0, 0, 0, 0, 0, 0) | 1291.4 [0.0 to 404404006.6] | 1997.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week.

5. Other Pre Specified Outcome: Anti-A-beta IgM (Immunoglobulin M) Titer at Specified Visits
Description: Geotmetric mean of anti-a-beta IgM titer from baseline of the preceding studies through the end of this study
Time Frame: Baseline of preceding studies to month 24 of this study (Week 210)
Population: The immunogenicity analysis population consisted of those in the safety analysis population who had baseline immunogenicity evaluation in the preceding study and at least one immunogenicity evaluation post injection. Since the study was early terminated and the data could not be obtained as planned, the IgM data were not summarized.
Arm/Group | 3 μg ACC-001+QS-21 | QS-21+(3 μg ACC-001+QS-21) | 10 μg ACC-001+QS-21 | 10 μg ACC-001+(10 μg ACC-001+QS-21) | QS-21+(10 μg ACC-001+QS-21) | PBS+(10 μg ACC-001+QS-21) | 30 μg ACC-001+QS-21 | 30 μg ACC-001+(30 μg ACC-001+QS-21) | QS-21+(30 μg ACC-001+QS-21) | PBS+(30 μg ACC-001+QS-21)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Other Pre Specified Outcome: The Mean Changes in Alzheimer's Disease Assessment Scale-Cognitive Behavior (ADAS-Cog) Score From Baseline at Week 26, 52, 78 and 104.
Description: The ADAS-Cog is a 12-item,objective measure of cognitive function, consisting of 1) Word Recall, 2) Naming Objects and Fingers, 3) Following Commands, 4) Constructional Praxis, 5) Ideational Praxis, 6) Orientation, 7) Word Recognition, 8) Recall of Test Instructions, 9) Spoken Language Ability, 10) Word-Finding Difficulty, 11) Comprehension of Spoken Language and 12) Concentration/Distractibility. For this study, the ADAS-Cog total score is derived by summing the individual scores from items 1 to 11, with higher scores indicating a greater degree of impairment. The total score ranges from 0 (no impairment) to 70 (worst impairment).
Time Frame: Baseline up to 24 Months
Population: The efficacy analysis population was all of the participants who received at least one injection in this study and had baseline efficacy evaluation in the preceding study and at least one efficacy evaluation post injection. Since the study was early terminated and the data could not be obtained as planned, the ADAS-Cog scores were not summarized.
Arm/Group | 3 μg ACC-001+QS-21 | QS-21+(3 μg ACC-001+QS-21) | 10 μg ACC-001+QS-21 | 10 μg ACC-001+(10 μg ACC-001+QS-21) | QS-21+(10 μg ACC-001+QS-21) | PBS+(10 μg ACC-001+QS-21) | 30 μg ACC-001+QS-21 | 30 μg ACC-001+(30 μg ACC-001+QS-21) | QS-21+(30 μg ACC-001+QS-21) | PBS+(30 μg ACC-001+QS-21)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Other Pre Specified Outcome: The Mean Changes in Disability Assessment for Dementia (DAD) Score From Baseline at Week 26, 52,78 and 104.
Description: The DAD is administered through an interview with the caregiver and measures instrumental and basic activities of daily living. A total score is obtained by adding the rating for each question and converting this total score out of 100. Higher scores represent less disability in ADL while lower scores indicate more dysfunction.
Time Frame: Baseline up to 24 Months
Population: The efficacy analysis population was all of the participants who received at least one injection in this study and had baseline efficacy evaluation in the preceding study and at least one efficacy evaluation post injection. Since the study was early terminated and the data could not be obtained as planned, the DAD scores were not summarized.
Arm/Group | 3 μg ACC-001+QS-21 | QS-21+(3 μg ACC-001+QS-21) | 10 μg ACC-001+QS-21 | 10 μg ACC-001+(10 μg ACC-001+QS-21) | QS-21+(10 μg ACC-001+QS-21) | PBS+(10 μg ACC-001+QS-21) | 30 μg ACC-001+QS-21 | 30 μg ACC-001+(30 μg ACC-001+QS-21) | QS-21+(30 μg ACC-001+QS-21) | PBS+(30 μg ACC-001+QS-21)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Other Pre Specified Outcome: The Mean Changes in Neuropsychological Test Battery (NTB) Score From Baseline at Week 26, 52, 78 and 104.
Description: The NTB is a composite of nine widely used neuropsychological tests that assess immediate and delayed recall of verbal and visual information, attention, verbal fluency and executive function. The cognitive tests included in the NTB are the Wechsler Memory Scale (WMS) Visual-Paired Associates (immediate and delayed), WMS-Verbal Paired Associates (immediate and delayed), Rey Auditory Verbal Learning Test (immediate and delayed), WMS-Digit Span, Controlled Word Association Test, and Category Fluency Test. The NTB z-score is used for analysis. The z-score for each component is calculated through the following formula: z = (y_visit - y_base)/SD_base, where y_visit is a value at a particular time point and y_base is the average test score, and SD_base is the SD based on all participants' observed baseline scores in the study.
Time Frame: Baseline up to 24 Months
Population: The efficacy analysis population was all of the participants who received at least one injection in this study and had baseline efficacy evaluation in the preceding study and at least one efficacy evaluation post injection. Since the study was early terminated and the data could not be obtained as planned, the NTB scores were not summarized.
Arm/Group | 3 μg ACC-001+QS-21 | QS-21+(3 μg ACC-001+QS-21) | 10 μg ACC-001+QS-21 | 10 μg ACC-001+(10 μg ACC-001+QS-21) | QS-21+(10 μg ACC-001+QS-21) | PBS+(10 μg ACC-001+QS-21) | 30 μg ACC-001+QS-21 | 30 μg ACC-001+(30 μg ACC-001+QS-21) | QS-21+(30 μg ACC-001+QS-21) | PBS+(30 μg ACC-001+QS-21)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Other Pre Specified Outcome: The Mean Changes in Mini-Mental State Examination (MMSE) Score From Baseline at Week 12, 26, 36, 52, 66, 78, 91 and 104.
Description: The MMSE is a brief, structured examination of cognitive function. It has a total score of 30 points, and any score equal to or lower than 26 points indicates cognitive impairment.
Time Frame: Baseline up to 24 Months
Population: The efficacy analysis population was all of the participants who received at least one injection in this study and had baseline efficacy evaluation in the preceding study and at least one efficacy evaluation post injection. Since the study was early terminated and the data could not be obtained as planned, the MMSE scores were not summarized.
Arm/Group | 3 μg ACC-001+QS-21 | QS-21+(3 μg ACC-001+QS-21) | 10 μg ACC-001+QS-21 | 10 μg ACC-001+(10 μg ACC-001+QS-21) | QS-21+(10 μg ACC-001+QS-21) | PBS+(10 μg ACC-001+QS-21) | 30 μg ACC-001+QS-21 | 30 μg ACC-001+(30 μg ACC-001+QS-21) | QS-21+(30 μg ACC-001+QS-21) | PBS+(30 μg ACC-001+QS-21)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- 3μg ACC-001 Treat: A group of participants who received IM injection of active vaccine ACC-001 (3 μg) + adjuvant QS-21 (50 μg) both in the preceding studies and in this study (Day 1, month 6, 12, and 18)
- 3μg Control: A group of participants who received IM injection of adjuvant QS-21 (50 μg) in the preceding studies and acctive vaccine ACC-001 (3 μg) + adjuvant QS-21 (50 μg) in this study (Day 1, month 6, 12, and 18)
- 10ug ACC-001 Treat: A group of participants who received IM injection of active vaccine ACC-001 (10 μg) with or without adjuvant QS-21 (50 μg) in the preceding studies and ACC-001 (10 μg) + adjuvant QS-21 (50 μg) in this study (Day 1, month 6, 12, and 18)
- 10μg Control: A group of participants who received IM injection of adjuvant QS-21 (50 μg) or PBS in the preceding studies and active vaccine ACC-001(10 μg) + adjuvant QS-21 (50 μg) in this study (Day 1, month 6, 12, and 18)
- 30μg ACC-001 Treat: A group of participants who received IM injection of active vaccine ACC-001 (30 μg) with or without adjuvant QS-21 (50 μg) in the preceding studies and ACC-001 (30 μg) + adjuvant QS-21 (50 μg) in this study (Day 1, month 6, 12, and 18)
- 30μg Control: A group of participants who received IM injection of adjuvant QS-21(50 μg) or PBS in the preceding studies and active vaccine ACC-001 (30 μg) + adjuvant QS-21 (50 μg) in this study (Day 1, month 6, 12, and 18)
- Total: All participants
Arm/Group | 3μg ACC-001 Treat | 3μg Control | 10ug ACC-001 Treat | 10μg Control | 30μg ACC-001 Treat | 30μg Control | Total
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/3 | 7/17 | 1/7 | 2/13 | 0/6 | 10/53
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3 | 15/17 | 5/7 | 10/13 | 6/6 | 46/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3μg ACC-001 Treat (N=7) | 3μg Control (N=3) | 10ug ACC-001 Treat (N=17) | 10μg Control (N=7) | 30μg ACC-001 Treat (N=13) | 30μg Control (N=6) | Total (N=53)
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Polychondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cerebral atrophy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Impulsive behaviour (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3μg ACC-001 Treat (N=7) | 3μg Control (N=3) | 10ug ACC-001 Treat (N=17) | 10μg Control (N=7) | 30μg ACC-001 Treat (N=13) | 30μg Control (N=6) | Total (N=53)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Glaucoma (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2
Dental caries (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 3
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Eructation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2
Rectal prolapse (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 2 | 1 | 2 | 2 | 2 | 2 | 11
Injection site haemorrhage (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Injection site nodule (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 1 | 2 | 1 | 2 | 2 | 1 | 9
Injection site pruritus (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Injection site swelling (General disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 4
Irritability (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Puncture site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 4
Biliary cirrhosis primary (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Balanitis candida (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 2
Nasopharyngitis (Infections and infestations) | 1 | 1 | 4 | 2 | 3 | 1 | 12
Periodontitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 0 | 0 | 1 | 5
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 2
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lymphocyte morphology abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Metamyelocyte percentage increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Protein urine present (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 1 | 1 | 5
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Apraxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cerebral microhaemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cerebral ventricle dilatation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 3
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Intercostal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lacunar infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 2
Occipital neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Visual field defect (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Intentional self-injury (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Logorrhoea (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Enuresis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 3

LIMITATIONS AND CAVEATS:
Since the study was early terminated and the data could not be obtained as planned, only part of the immunogenicity and safety results were summarized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.